CLINICAL TRIAL: NCT04237909
Title: Effects of Intraovarian Injection of Autologous Platelet Rich Plasma on Ovarian Reserve and IVF Outcome Parameters in Women With Premature Ovarian Insufficiency and Poor Ovarian Response
Brief Title: Effects of Intraovarian Platelet Rich Plasma in Women With Poor Ovarian Response and Premature Ovarian Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Bulent Tiras, Prof., Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATADEK 2019/8-18
Record Dates: First submitted 2020-01-12; First posted 2020-01-23 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Premature Ovarian Failure; Diminished Ovarian Reserve
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: After the couples are recruited for the study, Antral follicle count (AFC), serum anti-mullerian hormone (AMH) and follicle stimulating hormone (FSH) levels will be determined at baseline and will be repeated beginning with the first menstrual cycle. Approximately 20 ml of blood sample will be collected under sterile conditions, and PRP will be prepared. The same day, within 2 hours of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into at least one ovary Ovarian reserve (AFC, FSH, AMH), and IVF laboratory outcome parameters (number of MII oocytes, 2PN embryos, cleavage stage embryos) will be followed for six sequential months. Spontaneous pregnancies will also be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian Reserve (Experimental): Patients with diminished ovarian reserve or premature ovarian insufficiency
  Interventions: Biological: PRP injection into at least one ovary

INTERVENTIONS:
Biological: PRP injection into at least one ovary — The same day, within 2 hours of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into at least one ovary using a 35 cm 17 G single lumen needle. The injection will be done underneath the ovarian cortex to the subcortical and stromal areas. Approximately 2-4cc of the PRP solution will be injected into each ovary. After the procedure, the patients will be taken to the recovery room and will be observed for 30-40 minutes and also be discharged home on the same day.

SUMMARY:
Reproductive age women diagnosed with poor ovarian response (POR) based on Poseidon criteria and premature ovarian insufficiency (POI) based on ESHRE criteria and with a history of at least one prior failed IVF cycle will be recruited for the study. Antral follicle count (AFC), serum anti-mullerian hormone (AMH), and early follicular phase serum follicle stimulating hormone (FSH) levels will determined at baseline. Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols and will be injected to at least one ovary. Ovarian reserve parameters and IVF outcomes will be determined.

DETAILED DESCRIPTION:
Reproductive age women diagnosed with POR based on Poseidon criteria and POI based on European Society of Human Reproduction and Endocrinology (ESHRE) criteria with a history of at least one prior failed IVF cycle will recruited for the study. Antral follicle count (AFC), serum anti-mullerian hormone (AMH), and early follicular phase serum follicle stimulating hormone (FSH) levels will be determined at baseline. Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols. PRP injection will be performed under sedation anesthesia, using a 35 cm 17 G needle under transvaginal ultrasound guidance. On the 2-4th days of the first six menstrual cycles following the procedure, AFC, AMH, and FSH levels will be re-assessed. Patients with at least one antral follicle will be started on ovarian stimulation for in-vitro fertilization- intracytoplasmic sperm injection (IVF-ICSI), followed by embryo banking/ preimplantation genetic testing- aneuploidy (PGT-A) or embryo transfer. Markers of ovarian reserve (AFC, FSH, AMH), and IVF laboratory outcome parameters (number of metaphase II (MII) oocytes, 2PN(pronucleus) embryos, cleavage stage, blastocyst embryos) will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of >1 year infertility duration with at least one ovary, who fulfilled the ESHRE criteria,
* Patients diagnosed with POR based on Poseidon criteria and with a history of at least one prior failed IVF cycle

Exclusion Criteria:

* Presence of pregnancy,
* previous diagnosis of any malignancy,
* ovarian insufficiency secondary to sex chromosome etiology,
* prior major lower abdominal surgery resulting in pelvic adhesions,
* anticoagulant use for which plasma infusion is contraindicated,
* current or previous (Immunoglobulin A (IgA) deficiency

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve parameters | 6 months
  Number of participants with intraovarian injection of autologous PRP as assessed by blood hormone analysis and ultrasonographic antral follicle counts, change in serum FSH, AMH levels and number of antral follicle counts.

SECONDARY OUTCOMES:
Ovarian response to stimulation | 12 months
  Number of participants with intraovarian injection of autologous PRP as assessed by number antral follicle counts on ultrasound, eggs, and embryos in the laboratory, change from baseline in number of developing follicles, and percentage of obtained eggs and fertilized embryos.

OTHER OUTCOMES:
IVF outcomes | 15 months
  Number of participants with ovarian PRP as assessed by number of clinical pregnancies, change in the percentage of clinical pregnancy rates with IVF treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yigit Cakiroglu, Assoc.Prof., Study Director — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Result] Leijdekkers JA, Eijkemans MJC, van Tilborg TC, Oudshoorn SC, van Golde RJT, Hoek A, Lambalk CB, de Bruin JP, Fleischer K, Mochtar MH, Kuchenbecker WKH, Laven JSE, Mol BWJ, Torrance HL, Broekmans FJM; OPTIMIST study group. Cumulative live birth rates in low-prognosis women. Hum Reprod. 2019 Jun 4;34(6):1030-1041. doi: 10.1093/humrep/dez051. PMID 31125412
- [Result] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Result] Sfakianoudis K, Simopoulou M, Nitsos N, Lazaros L, Rapani A, Pantou A, Koutsilieris M, Nikas Y, Pantos K. Successful Implantation and Live Birth Following Autologous Platelet-rich Plasma Treatment for a Patient with Recurrent Implantation Failure and Chronic Endometritis. In Vivo. 2019 Mar-Apr;33(2):515-521. doi: 10.21873/invivo.11504. PMID 30804135